CLINICAL TRIAL: NCT01135030
Title: Anterior Referencing Vs. Posterior Referencing in Minimally Invasive Total Knee Arthroplasty
Brief Title: Anterior Referencing Versus Posterior Referencing in Minimally Invasive Total Knee Arthroplasty
Acronym: AR vs PR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heekin Orthopedic Research Institute (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Principal Investigator, R. David Heekin, R. David Heekin, M.D., Heekin Orthopedic Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-09-03
Record Dates: First submitted 2010-05-26; First posted 2010-06-02 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Osteoarthritis
Keywords: total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posterior referencing (Active Comparator)
  Interventions: Procedure: Total knee
- Anterior referencing (Active Comparator)
  Interventions: Procedure: Total knee

INTERVENTIONS:
Procedure: Total knee — Primary Total knee

SUMMARY:
The purpose of this study is to look at two different referencing systems for total knee replacement surgery. In anterior referencing system, referencing cuts are made from the front surface of the femur. This allows for a more exact cut. The anterior referencing system is more difficult for the surgeon to use. This may increase surgery time. Posterior referencing, on the other hand, references cuts from the back of the femur. The posterior referencing system is quick and easy for the surgeon to use. Posterior referencing may lead to notching of the femur. The risk of notching is very low and may not affect your results. This is a study that has never been done before. Dr. Heekin uses both referencing systems in his practice. He would like to determine which knee referencing system allows for greater knee flexion after surgery. Knee flexion correlates with function and the ability to return to everyday activities. For example, getting up from a chair, going up and down stairs, stooping, and kneeling.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a male or non-pregnant female between the ages of 21-80.
2. Patient requires cemented primary total knee replacement.
3. Patient has a diagnosis of osteoarthritis (OA), traumatic arthritis (TA), or avascular necrosis (AVN).
4. Patient has intact collateral ligaments.
5. Patient has signed and dated an IRB approved study specific consent form.
6. Patient is able and willing to participate in the study according to the protocol for the full length of expected term of follow-up, and to follow their physician's directions.
7. Patient has failed to respond to conservative treatment modalities.
8. Patient's contralateral knee is without symptomatic degenerative disease.

Exclusion Criteria:

1. Patient has had a prior procedure of high tibial osteotomy, cruciate ligament reconstruction or patellectomy of the surgical knee.
2. Patient is morbidly obese (BMI >30).
3. Patient has a deformity at the involved knee greater than 45degrees of flexion, 45 degrees of varus or 45 degrees of valgus.
4. Patient has an active or suspected latent infection in or about the knee joint.
5. Patient has a malignancy in the area of the involved knee joint.
6. Patient has a diagnosed systematic disease that would affect the subject's welfare or overall outcome of the study (i.e. moderate to severe osteoporosis, Paget's disease, renal osteodystrophy) or is immunologically suppressed, or receiving steroids in excess of physiologic dose requirements.
7. Patient has a neurological deficit, which interferes with the patient's ability to limit weight bearing or places an extreme load on implant during the healing period.
8. Female patient is or plans to become pregnant during the course of the study.
9. Patient has a known sensitivity to device materials.
10. Patient has prior diagnosis of diabetic or peripheral neuropathy in operative extremity or other neurologic disease affecting limb strength (i.e. Polymyositis, multiple sclerosis).
11. Patient's bone stock is compromised by disease or infection, which cannot provide adequate support and/or fixation to the prosthesis.
12. Patient has a TKA on the contralateral side less than six months post-op.
13. Patient has participated in an orthopaedic clinical investigation involving the hip or knee joint in the last 12 months.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
greater flexion after surgery | 12 months

SECONDARY OUTCOMES:
greater flexion after surgery | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Heekin Orthopedic Specialists, Jacksonville, Florida, United States